CLINICAL TRIAL: NCT02544828
Title: Does Intraoperative Intravenous Iron Sucrose Enhance Postoperative Oxygenation Profile in Total Arthroplasty Surgery?
Brief Title: Intravenous Iron Sucrose in Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUH1160093
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; knee arthroplasty; iron
MeSH Terms: conditions — Osteoarthritis | interventions — Ferric Oxide, Saccharated; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Iron Sucrose 200mg
  Interventions: Drug: Iron Sucrose 200mg
- Control Group (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Iron Sucrose 200mg — Iron Sucrose 200mg is administered after anesthesia induction.
  Arms: Experimental group
Drug: placebo — placebo (normal saline) is administered after anesthesia induction
  Other Names: normal saline
  Arms: Control Group

SUMMARY:
The objective of the present study is to determine the impact of intraoperative IV-iron supplementation on postoperative oxygenation profile by comparing the postoperative PaO2/FiO2 ratio with or without IV-iron supplementation in old patients undergoing elective uni-limb arthroplasty surgery.

DETAILED DESCRIPTION:
Participation and recruitment: Patients undergoing elective total knee arthroplasty due to osteroarthritis will be interviewed for participation and recruited after providing written informed consent.

Randomization and group allocation:

All recruited patients will be given patient identification number (PIN) for the present study of 01-76 according to their order of interview and recruitment.

Investigators will prepare 33 yellow and 33 green cards, which will be inserted in 76 thick-paper envelopes. Then, all envelopes will be sealed, mixed and randomly allocated to get numbers of 01 to 76 (Envelop number).

After printing the envelope number outside envelope, all sealed envelopes with cards will be conveyed to and kept in pharmacy department.

Preparation and Administration of study drug:

Pharmacist will open the envelope with the number same to PIN and check the color of the card inside at study on operation day.

According to the color of the card, IV-iron or placebo will be prepared for the patient: IV-iron for yellow card; placebo for green cards, respectively.

The study drug will be covered by black-tape by pharmacist and delivered to the operation theater.

IV-iron or placebo will be infused through already established intravenous line within 30 min after anesthesia induction by attending anesthesiologist who is not aware of the patient's group-allocation.

Patient data and statistical analyses:

The information regarding the patient's group allocation will be kept in the pharmacy department till the end of the study and conveyed during the data analyses after completion of the 76th patient participation and discharge.

Patient's data PaO2, FiO2, Hb, intra-op and postop-transfusion amount, intraop- and postop-bleeding amount will be determined from the patients' medical record after patient's discharge.

All statistical analyses will be performed after the 76th patient's discharge and data acquisition.

Surgical procedures:

All surgical procedures will be performed using standardized institutional anesthetic and surgical protocols, antibiotic and antithrombotic prophylaxis, transfusion protocols, and post-operative analgesia.

All TKA will be performed using a pneumatic tourniquet, which is deflated after wound closure. Closed suction drains, which are removed on the second post-operative day, will be placed in all operations.

Transfusion protocol:

Following allogenic blood transfusion protocol will be uniformly applied by anesthesiologists and surgeons to all patients in the operating theater, the post-operative anesthesia care unit, and the ward for the entire duration of hospitalization: blood transfusion of packed RBC will not be performed unless patient's Hb level is < 9 g/dL without any signs and/or symptoms of acute anemia such as hypotension, tachycardia, tachypnea, dizziness, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis in knee joint undergoing elective uni-limb total knee arthroplasty surgery
* Patients provided a written informed consent.
* Patients with s-ferritin < 300 mg/dl (male) or 200 mg/dl (female)
* Patients with preoperative serum hemoglobin concentration >13 g/dL (male) and >12 g/dL (female)
* Patients with PaO2/FiO2 ratio >150

Exclusion Criteria:

* Patients with history of anaphylaxis, iron overload, active infection.
* Patients with endocrine disease
* Patients received or receiving intraoperative and preoperative blood salvaged, allogenic blood transfusion, anti-fibrinolytic agents or recombinant human erythropoietin, or undergoing acute normovolemic hemodilution.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 24 hour
  Intergroup-difference in PaO2/FiO2 ratio

SECONDARY OUTCOMES:
arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 2 hour
  intergroup-difference in PaO2/FiO2 ratio
arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 48 hour
  intergroup-difference in PaO2/FiO2 ratio
serum hemoglobin concentration | postoperative 2 hour
  serum hemoglobin concentration, g/dL
postoperative transfusion red blood cell amount | postoperative 24 hour
  postoperative transfusion of packed red blood cell, ml